CLINICAL TRIAL: NCT02150187
Title: Evaluation of the Efficacy of Hcap Formula Nutrition Supplement for Treatment of Men With Androgenic Alopecia: A Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Efficacy of Nutrition Supplement for Treatment of Men With Hair Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Family Marketing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ProHair01
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia; Male; Baldness; hair loss pattern
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCap Formula (Experimental): Pill of HCap Formula every other day for 6 month during the treatment phase; Follow up phase: nothing.
  Interventions: Dietary Supplement: HCap Formula
- Placebo (Placebo Comparator): Same as treatment with placebo pills
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HCap Formula — Pill should be taken every other day during the treatment phase.
  Arms: HCap Formula
Dietary Supplement: Placebo — Similar pills without active ingredients
  Arms: Placebo

SUMMARY:
HCap Formula is composed of medicinal plants, vitamins and minerals. The purpose of this study is to evaluate the efficacy of HCap Formula, a nutrition supplement for promoting hair growth in men with tendencies for hair loss.

DETAILED DESCRIPTION:
This study consists of a treatment phase (6 months) and a follow-up phase (6 month ). Eligible subjects will be randomly assigned to receive treatment with the study medication or placebo. Subjects will visit the clinic at 3, 6, and 12 months after treatment start for safety and efficacy evaluations.

HCap Formula or placebo tablets will be taken orally every other day during 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between 18-40 years of age.
2. No abnormality in blood tests analysis
3. Present with mild to moderate androgenic alopecia (AGA) graded IIv, IIIv, IV or V according to the Hamilton-Norwood classification
4. Willingness to use the same shampoo, refrain from change in hair style, and refrain from hair dyeing during the study.
5. Willingness to refrain from any therapy affecting hair during the study
6. Willingness to have photographs of the treated area taken.
7. Willingness to follow the treatment schedule and post treatment follow-up.
8. Willingness not participate on other studies during the study course

Exclusion Criteria:

General

1. Having a known allergy to any of the ingredients in the test products;
2. Participation in a study of another device or drug within one month prior to enrollment or during the study.

   Hair treatments/ scalp condition
3. Undergone hair transplant surgery, scalp reduction surgery
4. Having hair weave or tattooing of the alopecic area.
5. Other hair loss disorders, such as alopecia areata, scarring alopecia.
6. Suffering from any active dermatological condition in the treated area such as scalp atrophy, which in the opinion of the investigator might interfere with clinical evaluation.

   Medications

   Use of the following medications within the past 6 months:
7. Prescription or over-the-counter systemic or topical treatment specific for androgenic alopecia (such as minoxidil, finasteride, dutasteride).
8. 5α-reductase inhibitors for prostate conditions (e.g. benign prostate hyperplasia, prostate cancer) and hormone replacement therapy for transgenders
9. Medications with anti-androgenic properties (cyproterone, spironolactone, ketoconazole, flutamide, progesterone, and bicalutamide)
10. Medications that can potentially cause hypertrichosis (e.g. cyclosporine, diazoxide, phenothiazines, zidovudine, tamoxifen, carpronium chloride),
11. Medications that can potentially cause alopecia such as oral glucocorticoids, lithium, phenothiazines, tamoxifen.

    Use of the following medications within the past 3 months:
12. Botanicals/nutraceuticals for hair growth
13. Steroids - systemic steroids for more than 14 days (e.g. corticosteroids, anabolic steroids) or topical steroids on the area of hair loss.

    Other medical conditions
14. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), uncontrolled hypertension, symptomatic hypotension, hyper/hypo thyroidism, or pertinent neurological disorders.
15. Suffering from serious medical condition that could adversely affect hair loss such as immunosuppression/immune deficiency disorders (including HIV), history of cancer or having/undergoing any form of treatment for active cancer, connective tissue disorder, inflammatory bowel disease
16. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in Terminal Hair Count at 26 Weeks Compared to Baseline | Baseline, 26 Weeks
  The primary outcome will be change in the terminal hair count from baseline to 26 Weeks within a 3 cm diameter circle based on macro-photographs of the same area. The treatment group will be compared to the control.

SECONDARY OUTCOMES:
Global Assessment of Improvement from Baseline to 26 and 52 weeks Assessed for Vertex and Frontal Views Separately | Baseline, 26 weeks, 52 weeks
  Assessment of improvement using a 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3). This assessment will be performed by comparing the global photographs obtained at Baseline with those subsequently obtained at baseline, 26, and 52 weeks. This assessment will be carried out separately on the global photography of the vertex and frontal views

CONTACTS AND LOCATIONS:
Overall Officials: David J Friedman, MD, Principal Investigator — Friedman Skin & Laser Center; Lilach Gavish, PhD, Study Director — Friedman Skin & Laser Center
Locations (1):
- Dr David Friedman Laser & Skin Center, Jerusalem, Israel